CLINICAL TRIAL: NCT01164553
Title: A Randomized, Double-Blind, Phase I Study Comparing an Increased Dose(s) (0.5 ml) of Trivalent Inactivated Influenza Vaccine (TIV) With Standard Dose(s) (0.25 ml) TIV in Children 6-35 Months of Age
Brief Title: Comparison of Flu Vaccine Doses in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 09-0018; N01AI80006C
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2012-10

CONDITIONS: Influenza
Keywords: influenza, pediatric, vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Group 2, 0.5 mL TIV (Experimental): Naive cohort participants (n=180) receive 0.25 mLTrivalent Inactivated Vaccine (TIV) in two intramuscular doses 28-42 days apart. Fully Primed cohort participants (previously vaccinated) (n=40) will receive 0.5 mL Trivalent Inactivated Influenza Vaccine (TIV) in one intramuscular dose.
  Interventions: Biological: Trivalent Inactivated Influenza Vaccine
- Group 1, 0.25 mL TIV (Active Comparator): Naive cohort participants (n=90) receive 0.25 mLTrivalent Inactivated Vaccine (TIV) in two intramuscular doses 28-42 days apart. Fully Primed cohort participants (previously vaccinated) (n=20) will receive 0.25 mL Trivalent Inactivated Influenza Vaccine (TIV) in one intramuscular dose
  Interventions: Biological: Trivalent Inactivated Influenza Vaccine

INTERVENTIONS:
Biological: Trivalent Inactivated Influenza Vaccine — Either a standard pediatric dose (0.25 ml) or a larger dose (0.5 ml) of Trivalent Inactivated Influenza Vaccine (TIV) (Fluzone®) administered intramuscularly (IM) in the thigh with a 25 gauge 1 inch needle. Naive cohort (enrolled over two influenza seasons (2010-11 and 2011-12)) will receive vaccine in two IM doses 28-42 days apart, Fully Primed cohort (enrolled in one influenza season (2010-11)) will receive vaccine in one IM dose.

SUMMARY:
The purpose of this study is to evaluate the possibility that giving an increased dose of flu vaccine to children 6 through 35 months of age will improve protection against influenza without increasing side effects. Investigators will evaluate the body's response to the vaccine. Male and female participants' ages 6-35 months, who have never received flu vaccine, and those ages 12-35 months, who have been previously vaccinated, will participate in the study for about 7 months. Vaccine naïve study participants will receive two doses of flu vaccine, either the 0.25 mL dose (Group 1) or 0.5 mL dose (Group 2). Previously vaccinated subjects will receive one dose of flu vaccine, either the 0.25 mL dose (Group 1) or 0.5 mL dose (Group 2). Study procedures include physical examination, memory aids, blood sampling and a follow-up phone call about 6 months after the last vaccine dose.

DETAILED DESCRIPTION:
Influenza is an important cause of morbidity and mortality among both children and adults. Influenza A and/or B viruses cause yearly epidemics in the United States with an average of 36,000 deaths and 114,000 hospitalizations annually. Children have the highest rates of infection. Influenza is also associated with substantial numbers of hospitalizations among young infants. Because of the limited data available and the variability of reported seroresponses to doses of 0.25 ml in children 6-35 months of age, investigators hypothesize that a higher dose will be more consistently immunogenic. In addition, since currently licensed trivalent inactivated influenza (TIV) vaccines are well tolerated with minimal systemic and local adverse events, investigators hypothesize that administering a higher dose of 0.5 ml to this age group will be well-tolerated. Therefore, investigators propose to compare the safety and immunogenicity of 0.25 ml doses of TIV to that of 0.5 ml doses of TIV when administered to children 6-35 months of age. The proposed study is a phase I, two-arm, 1:2 randomized, double-blinded trial comparing the safety and immunogenicity of increased dose(s) (0.5 ml) with standard dose (0.25 ml) of TIV in children 6-35 months of age with and without a history of previous TIV vaccination. The population will include a Naïve Cohort: 270 healthy male and female children who are 6-35 months of age and have never received an influenza vaccination; and a Fully Primed Cohort: 60 healthy male and female children who are 12-35 months of age and have received two doses of 2009-2010 H1N1 and two doses of TIV at anytime in the past as defined for purposes of this study. Either a standard pediatric dose (0.25 ml) or a larger dose (0.5 ml) of TIV will be administered intramuscularly in the anterolateral thigh with a 25 gauge 1" needle. The primary objective is to evaluate the safety of administering an increased dose(s) (0.5 ml) of TIV to children 6-35 months of age as compared to standard dose(s) (0.25 ml) of TIV. The secondary objective is to compare the humoral immune responses to TIV antigens in children 6-35 months of age who receive the increased dose(s) of TIV to those who receive the standard dose(s) of TIV.

ELIGIBILITY:
Inclusion Criteria:

All Subjects

* Healthy children 6-35 months of age (naïve cohort) or 12-35 months of age (fully primed cohort)
* Free of obvious health problems as established by medical history and clinical examination before entering the study
* Parent/legal guardian willing and capable of signing written informed consent
* Parent/legal guardian expected to be available for entire study
* Parent/legal guardian can be reached by telephone

Fully Primed Cohort

-Have received two doses of 2009-2010 H1N1 and two doses of trivalent inactivated influenza vaccine (TIV) at anytime in the past as defined for the purpose of this study.

Exclusion Criteria:

All Subjects:

* Have known allergy to eggs or other components of the vaccine. *Refer to the Fluzone package insert for a list of vaccine components.
* Known or suspected latex allergy.
* Former premature infants (<32 weeks).
* History of bronchodilator use more than 2 times per week within 28 days of vaccination.
* Significant underlying chronic illness (e.g., congenital heart disease, bronchopulmonary dysplasia).
* Immunodeficiency disease or use of immunosuppressive therapy by the participant, including perinatal exposure to or infection with human immunodeficiency virus (HIV), or known infection with hepatitis B or hepatitis C.
* Any other condition that, in the clinical judgment of the investigator, may interfere with vaccine evaluation. Children receiving antibiotics are eligible for enrollment.
* Have long term use of glucocorticoids including oral, parenteral or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months. (Nasal and topical steroids are allowed.)
* Previous, exposure to an investigational drug or investigational vaccine within 28 days prior to vaccination in this trial.
* Plans for participation in another clinical trial with an investigational drug or investigational vaccine for the duration of this study.
* History of Guillain-Barré syndrome or any other neuromuscular disease.
* History of seizures (including febrile seizures).

Naïve Cohort:

* Any prior influenza vaccination.
* History of documented laboratory-confirmed influenza infection.

Fully primed Cohort:

* Have not received two doses of 2009-2010 H1N1 and two doses of trivalent inactivated influenza vaccine (TIV) at anytime in the past as defined for the purpose of this study.
* Allergic response to prior receipt of influenza vaccine.

Criteria for temporarily delaying vaccine administration for both groups:

The following conditions are temporary or self-limiting and a subject may be included in the study once the condition(s) has/have resolved, provided that the subject is otherwise eligible:

* Receipt of blood products in the previous 90 days
* Fever (axillary temperature > 100.0 degrees Fahrenheit/37.8 degrees Celsius), or an acute illness within 48 hours of enrollment.
* Receipt of any live vaccines within four weeks or any inactivated vaccines within two weeks of study vaccination.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 243 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Incidence of local and systemic side effects in children receiving the standard dose (0.25ml) or increased dose (0.5 ml) of Trivalent Inactivated Influenza Vaccine. | In the week after each vaccination.
Incidence of adverse events in children receiving the standard dose (0.25ml) or increased dose (0.5 ml) of Trivalent Inactivated Influenza Vaccine (TIV). | In the 4 weeks after each vaccination.

SECONDARY OUTCOMES:
Percent of children who develop hemagglutinin inhibition (HAI) antibody titers greater than or equal to 1:40 (presumed protective titers) and the percent with 4-fold rises. | Approximately 30 days after one or two standard (0.25 ml) or increased (0.5 ml) doses of Trivalent Inactivated Influenza Vaccine (TIV) in fully primed and naive children.
Geometric mean titer (GMT) of the hemagglutinin inhibition (HAI) antibody responses to each of the components of the Trivalent Inactivated Influenza Vaccine (TIV). | Approximately 30 days after one or two standard (0.25 ml) or increased (0.5 ml) doses of Trivalent Inactivated Influenza Vaccine in fully primed and naïve children.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Emory Children's Center - Pediatric Infectious Diseases, Atlanta, Georgia
  - Emory University School of Medicine - Emory Children's Center - Pediatric Infectious Diseases, Atlanta, Georgia
  - University of Iowa - Infectious Disease Clinic, Iowa City, Iowa
  - University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio
  - Vanderbilt University - Pediatric - Infectious Diseases, Nashville, Tennessee